CLINICAL TRIAL: NCT02293330
Title: Continuous Infusion Versus Automated Intermittent Bolus of Levobupivacaine 0,1% in Ultrasound Guided Subparaneural Sciatic Nerve Catheters. A Prospective Double Blind Randomised Study.
Brief Title: Continuous Versus Automated Bolus Infusion in Sciatic Nerve Catheters
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Antwerp (Other)
Responsible Party: Principal Investigator, Dr M. B. Breebaart, MD, University Hospital, Antwerp
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: 14/38/393
Record Dates: First submitted 2014-10-30; First posted 2014-11-18 (Estimated); Last update posted 2016-11-23 (Estimated); Status verified 2016-11

CONDITIONS: Hallux Valgus; Surgery
Keywords: continuous versus intermittent bolus sciatic nerve block
MeSH Terms: conditions — Hallux Valgus | interventions — Levobupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- C group (Experimental): continuous infusion of levobupivacaine
  Interventions: Drug: continuous infusion of levobupivacaine
- B group (Experimental): Intermittent bolus infusion of levobupivacaine
  Interventions: Drug: Intermittent bolus infusion of levobupivacaine

INTERVENTIONS:
Drug: continuous infusion of levobupivacaine — continuous infusion of levobupivacaine 0,125% at 5 ml/h , bolus dose 6 ml, lock out 30 minutes 4 hours limit: 60 ml/h
  Other Names: chirocaine
  Arms: C group
Drug: Intermittent bolus infusion of levobupivacaine — Intermittent bolus of levobupivacaine 0,125%: 0.1 ml /h and 9,8 ml bolus every two hours. Optional patient controlled bolus dose 6 ml, lock out 30 minutes, 4 hours limit: 60 ml/h
  Other Names: chirocaine
  Arms: B group

SUMMARY:
This study is developed to determine if the local anaesthetic dose can be reduced by the use of intermittent bolus technique compared to continuous infusion when the nerve catheter is placed underneath the paraneurium by ultrasound guidance in the popliteal fossa. Our primary outcome is local anesthetic use the first 48 hours after connecting the peripheral nerve catheter. Our hypothesis is that with an intermittent bolus less local anaesthetic is necessary the first postoperative 48 hours after surgery for adequate postoperative analgesia. As secondary outcomes the investigators study pain scores, motor block, sensory block, feeling of numbness, patient satisfaction, sleep quality and rescue analgesia during the nerve block and afterwards.

DETAILED DESCRIPTION:
Patients scheduled for foot surgery under general anaesthesia and a popliteal nerve catheter will be asked to take part and give informed consent. The anaesthesiologist performing the block, the patient and the independent observer will be blinded to the study group and the settings of the pump (CADD®-Solis) will be regulated and the data collected after 48 hours by an independent pain nurse or anaesthetist who is aware of the study group but does not register any other parameters.

Patients will be randomised by a computer-generated sequence, concealed by sealed envelopes. The envelope will be opened and the pump prepared by an independent pain nurse or anaesthesiologist who will not participate in registration of the parameters except extracting information out of the pump when the catheter is removed.

We expect to detect a 20 % increase in local anaesthetic dose for the continuous administration group (230 mg/48 hour). We used a standard deviation of 25%(58 mg) from a previous study. The minimum sample size required is 20 patients per group for a power of 80% with a 2-tailed significance level of 5%. We decided to include 25 patients in each group.

Before surgery

An IV access and standard monitoring is used throughout the procedure. A pre puncture scan will be performed and an experienced anaesthesiologist will perform all blocks. The block is performed in the lateral decubitus with a 12-18 MHz (megahertz) linear probe (BK medical®) and a solo long needle-catheter set (Pajunk®,18 gauge needle, 20 gauge catheter). The nerve will be visualised in a short axis image and the puncture will be done out of plane. Confirmation of accurate needle tip position will be confirmed by injection of nacl 0,9% (sodium chloride) and the appearance of a "twin- or triple halo sign". After confirmation of correct needle tip position 15 ml levobupivacaine 0,25% (chirocaine® Abbot)will be injected in between de peroneal and tibial nerve as an initial bolus. After injection a will be advanced 4 cm beyond the needle tip.

Correct catheter placement will be confirmed by ultrasound. A detailed description of block performance will be registered according to our standard hospital policy. The sensory block of the peroneal and tibial nerve will be separately tested by loss of cold sensation before transfer to the operating room, at least 20 minutes after the initial injection of lidocaine. When no block is detected it is considered as a block failure and the patient will be excluded from the study.

After performing the popliteal block the patients will be transferred to the operating room and receive general anaesthesia by an independent anaesthesiologist. Surgery will be performed with a tourniquet at 300 mm Hg. Standard monitoring is used during surgery (ecg, pulse oximetry and non invasive blood pressure measurement). Duration of surgery will be registered.

After the operation the patient will be transferred to the recovery room. Here the popliteal catheter will be connected pain pump (which will be defined as t=0) with an infusion protocol according to the study group:

C group: continuous infusion of levobupivacaine 0,125% (chirocaine ®, Abbot) B group: Intermittent bolus of levobupivacaine 0,125 ( chirocaine®Abbot) Both groups will have the possibility of administering a pca (patient controlled analgesia) bolus of 6 ml.

The Pump (CADD®-Solis Smiths medical) which will be started in the recovery room by an independent pain nurse or anaesthetist who is aware of the appointed study group (C group or B group). Pain scores ,motor block,sensory block and presence of numbness will be registered when the patient is awake enough to evaluate these parameters.

The patient will then be transferred to the ward after clear instructions of how to use the pain pump.The study will continue until 48 hours after starting the pump. Pain scores will be registered every four hours at the ward as well as feeling of numbness and sleep quality at regular intervals. During night hours (00-06)when the patient is sleeping pain scores will be registered as "S".When pain control is insufficient at the PACU or on the ward patients will receive paracetamol 1gr IV(Paracetamol® )and ketorolac (taradyal®) 30 mg IV. Tramadol ( contramal ®) 2 mg/kg will be given as rescue analgesia. On day one rescue analgesia will be provided orally .

All rescue analgesia or other medication will be registered.

48 hours after starting the pain pump the pump will be removed and all data will be collected and filed by an independent pain nurse or anaesthetist. This file will consist of a detailed description of the history of local anaesthetic administered, including total anaesthetic dose at 6,12,24 and 48 hours , frequency of extra boluses required and time intervals.

Before removing the nerve catheter the depth of the catheter is checked and bolus of nacl will be infused under ultrasound guidance and if possible correct placement can be confirmed after two days. Then the catheter will be removed.

After stopping the pump the patient will be asked if he or she was satisfied by the postoperative analgesic technique:

1. Satisfied
2. Sufficient
3. Not satisfied

The patient is discharged but is asked to register the exact time point when sensation and motor function (when a motor block was present) after catheter removal appeared. The patient will be called two days after discharge to register these parameters.

ELIGIBILITY:
Inclusion Criteria:

* scheduled for for surgery for hallux valgus pathology with general anesthesia and a popliteal nerve catheter (=sciatic nerve block)

Exclusion Criteria:

* neuromuscular disease,
* chronic pain,
* peripheral neuropathy in lower limb,
* contraindication for popliteal nerve block,
* unable to use pca (patient controlled analgesia),
* patient refusal

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2014-11; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
local anesthetic dose in 48 hours | 48 hours
  the total amount of local anesthetic dose (mg) in total administered by the pump connected to the sciatic nerve catheter from start of the pump until stop ( 48 hours after start)

SECONDARY OUTCOMES:
pains scores | 48 hours
  pain scores on a numeric rating scale (0-10) will b scored on regular intervals ( every 4 hours)
motor block (possibility of tow movement ( yes/no) | 48 hours
  possibility of tow movement ( yes/no) 6,12,24,30,36 and 48 hours after starting the pump)
sensory block loss of cold sensation (yes/no) | 48 hours
  loss of cold sensation ( yes/no) in peroneal an tibial dermatome , measured at 6,12,24,30,36 hours after starting the pump
numbness (sensation of numbness (0 = no, 1= yes but not disturbing, 2= yes and disturbing) | 48 hours
  sensation of numbness (0 = no, 1= yes but not disturbing, 2= yes and disturbing) measured at 6,12,24,30,36,48 hours after starting the pump
patient satisfaction 9satisfaction on a 10 point scal ( 0= very dissatisfied, 10 = very satisfied) | 48 hours
  satisfaction on a 10 point scal ( 0= very dissatisfied, 10 = very satisfied)

OTHER OUTCOMES:
first sensation after stopping the pomp | two days after discharge
  the patient is asked to note the time point (day, hour) at which sensation and /or motor function returned. A nurse will call two days after discharge to ask.

CONTACTS AND LOCATIONS:
Overall Officials: Margaretha Breebaart, Principal Investigator — University Hospital, Antwerp
Locations (1):
- University Hospital Antwerp, Antwerp, Belgium